CLINICAL TRIAL: NCT02514902
Title: Stroke and Traumatic Acute Brain Injury Line Indicator System for Emergent Recognition (STABILISER-I)
Acronym: STABILISER-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justin Fraser (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Justin Fraser, Asst Professor of Cerebrovascular, Endovascular, and Skull Base Surgery, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15-0166-F6A; NIH UL1TR000117 (Other: University of Kentucky CCTS High Impact Award)
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke; Traumatic Brain Injury
Keywords: Lateral Flow Device (LFD); Acute Stroke; Traumatic Brain Injury (TBI); Point of Care (POC); Biomarker
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lateral Flow Device (Experimental): Determine the feasibility of testing whole blood samples from patients with acute stroke (both ischemic and hemorrhagic) and traumatic brain injury being evaluated in the Emergency Department and Inpatient Services at University of Kentucky. No diagnostic or treatment decisions will be based on the results for any patient and the patient will not be told of the results.
  Interventions: Device: Lateral Flow Device

INTERVENTIONS:
Device: Lateral Flow Device — A drop of whole blood from a finger stick is placed on the lateral flow device at two different time points to indicate the presence of a neuronal specific biomarker. The results will also be correlated to severity of clinical and radiographic injury. Separate drops are evaluated similarly for serum levels. The objective is to determine feasibility of a diagnostic tool for stroke (ischemic and hemorrhagic and traumatic brain injury (TBI). No diagnostic results or resulting treatments will be applied to any subject.

SUMMARY:
In the search for a novel marker of stroke that could be rapidly assessed in blood, the investigators developed a point-of-care (POC) lateral flow device (LFD) that rapidly (< 15 min) detects levels of a biomarker that is released into blood following neuronal injury associated with stroke and traumatic brain injury. The protein's expression in human brain should serve as a useful biomarker of neuronal injury in stroke and traumatic brain injury.

DETAILED DESCRIPTION:
The use of a lateral flow device (LFD) to indicate the presence of a blood biomarker is feasible and may provide an important diagnostic tool for stroke and traumatic brain injury (TBI).

Primary Objectives:

1. Determine the first-in-humans feasibility using the investigators' biomarker lateral flow device on whole blood samples to diagnose patients with acute stroke (both ischemic and hemorrhagic) and traumatic brain injury being evaluated in the Emergency Department and Inpatient Services at University of Kentucky. Provide initial pilot data for estimating sensitivity and specificity of the assay.
2. Establish a visual ordinal grading scale that is easy to use clinically to judge the severity of injury, from the Lateral Flow Device result. Verify that the visual scale has inter-rater reliability, and evaluate it against a digital detection assay.
3. Examine the correlation between clinical and radiographic parameters of injury severity and blood levels of the biomarker. The investigators will correlate the results of the test with NIH Stroke Scale and with MRI infarct volume for ischemic stroke, with hemorrhage volume on CT for hemorrhagic stroke, and with Glasgow Coma Scale for Traumatic Brain Injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21-85 years old, male or female.
2. Suspected TBI, acute ischemic stroke, or nontraumatic/nonlesional intracerebral hemorrhage (ICH) based on clinical and radiographic evidence as determined and documented by the appropriate service (Trauma Service or Neurosurgery Service for TBI; Neurology or Neurosurgery Service for Stroke) at University of Kentucky.
3. Patients with impaired capacity may be included; as the pathology to be studied (stroke or TBI) may impair their capacity (please see attached required documentation regarding impaired capacity).

Exclusion Criteria:

1. Pregnant women as the effect of pregnancy on the biomarker testing result is as yet unknown.
2. While patients may be included with the above listed diagnoses, they may be excluded later if an alternate unlisted diagnosis is found to be the root cause of their presentation. An example would be a patient initially thought to have a stroke, who is discovered to be suffering from a seizure instead.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Whole Blood Biomarker Results on the Visual Analog Scale | Within 8 hours of time of injury/onset of stroke symptoms.
  Degree of response to a protein specific biomarker in whole blood as indicated by the Lateral Flow Device's analog scale: negative / mild / moderate / severe.

SECONDARY OUTCOMES:
Whole Blood Biomarker Results on the Visual Analog Scale | Within 48 ± 8 hours of time of injury/onset of stroke symptoms.
  Degree of response to a protein specific biomarker in whole blood as indicated by the Lateral Flow Device's analog scale: negative / mild / moderate / severe.
Serum Biomarker Results on the Visual Analog Scale | Within 8 hours of time of injury/onset of stroke symptoms.
  Degree of response to a protein specific biomarker in serum as indicated by the Lateral Flow Device's analog scale: negative / mild / moderate / severe.
Serum Biomarker Results on the Visual Analog Scale | Within 48 ± 8 hours of time of injury/onset of stroke symptoms.
  Degree of response to a protein specific biomarker in serum as indicated by the Lateral Flow Device's analog scale: negative / mild / moderate / severe.

CONTACTS AND LOCATIONS:
Overall Officials: Justin F. Fraser, MD, Principal Investigator — University of Kentucky Department of Neurological Surgery
Locations (1):
- University of Kentucky Deparment of Neurosurgery, UK Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No